CLINICAL TRIAL: NCT00616733
Title: An Open-label, Escalating-dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral CS-0777, Administered for 12 Weeks, in Patients With Multiple Sclerosis
Brief Title: 12-week Safety Evaluation of Oral CS-0777 in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: James Moberly, PhD, Senior Director, Clinical Development, Daiichi Sankyo, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS0777-A-U102; IND 77,409
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis, relapsing, secondary progressive, clinically isolated syndrome, MRI
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — CS 0777

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: CS-0777 tablets
- 2 (Experimental)
  Interventions: Drug: CS-0777 tablets
- 3 (Experimental)
  Interventions: Drug: CS-0777 tablets

INTERVENTIONS:
Drug: CS-0777 tablets — 0.1 mg, once-weekly, for 12 weeks
  Arms: 1
Drug: CS-0777 tablets — 0.3 mg, once-weekly or once every 2 weeks, for 12 weeks
  Arms: 2
Drug: CS-0777 tablets — 0.6 mg, once-weekly or once every 2 weeks, for 12 weeks
  Arms: 3

SUMMARY:
This is a 12-week study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of oral CS-0777 in patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of clinically isolated syndrome or a relapsing form(s) of MS, based on Poser or McDonald criteria (may include patients with secondary progressive disease)
* Clinical relapse within the past 3 years or a gadolinium enhancing lesion on a brain MRI scan within the past 12 months
* Baseline EDSS score of 0 - 6.5
* Female subjects who are sexually active, unless sterile or post-menopausal for at least 1 year, must be willing to use double-barrier contraception

Exclusion Criteria:

* Primary progressive MS
* Any medical condition that predisposes to immunocompromise
* History of malignancy, tuberculosis, invasive fungal infections, herpes zoster infection (or shingles), or other opportunistic infection, or any current active infection
* Concurrent diagnosis of any other autoimmune disease (eg, rheumatoid arthritis or lupus)
* Treatment with cyclophosphamide or mitoxantrone within 6 months of study initiation
* Treatment with cyclosporine, azathioprine, methotrexate or other immunosuppressant within 3 months of study initiation
* Treatment with interferon beta or glatiramer acetate within 2 months of study initiation
* Prior treatment with natalizumab or rituximab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability. | 12 weeks, with 4 weeks to follow-up

SECONDARY OUTCOMES:
Pharmacodynamic response (lymphocyte counts Pharmacokinetics Exploratory efficacy based on brain MRI lesions) | 12 weeks, with 4 weeks to follow up.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Denver, Colorado
  - Port Orange, Florida
  - Lenexa, Kansas
  - Billings, Montana
  - Philadelphia, Pennsylvania